CLINICAL TRIAL: NCT03086122
Title: The Impact of Obstructive Sleep Apnea in Erectile Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Ferran Barbe, Head of Respiratory Medicine at Hospital Universitari Arnau de Vilanova, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nº80-Separ2011
Record Dates: First submitted 2017-03-12; First posted 2017-03-22 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA; Erectile Dysfunction; CPAP treatment; Endothelial Dysfunction; Cardiovascular risk
MeSH Terms: conditions — Sleep Apnea, Obstructive; Erectile Dysfunction | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Obstructive Sleep Apnea (OSA) (No Intervention): OSA patients without erectile dysfunction (ED).
- OSA + ED (No Intervention): OSA patients with erectile dysfunction diagnosis who are randomly allocated to not receive continuous positive airway pressure (CPAP).
- OSA + ED + CPAP (Experimental): OSA patients with erectile dysfunction diagnosis who are randomly allocated to receive CPAP.
  Interventions: Device: Continuous positive airway pressure

INTERVENTIONS:
Device: Continuous positive airway pressure — Continuous positive airway pressure treatment for patients randomized to CPAP treatment group. Treatment duration: 3 months.
  Other Names: CPAP
  Arms: OSA + ED + CPAP

SUMMARY:
The syndrome of obstructive sleep apnea (OSA) is a common condition that affects 2-4% of the general population, causing an increase in sympathetic activity, changes in systemic blood pressure, and is associated with cardiovascular disease. The pathophysiological mechanisms that are altered as a result of the events associated with obstructive sleep apnea (hypoxia-reoxygenation, arousals and sleep fragmentation), are associated with an increased risk of developing erectile dysfunction in patients with Obstructive Sleep Apnea. Until today, the studies linking Erectile Dysfunction with Obstructive Sleep Apnea (OSA) are epidemiological studies.

The alterations in the expression profile of endothelial and cardiovascular dysfunction biomarkers and sex hormones disorders that are altered as a result of the events associated with OSA are associated to erectile dysfunction development.

Treatment with continuous positive airway pressure (CPAP) reverses the effects of OSA and patients with erectile dysfunction may improve erectile function.

The primary objective of the study is:

1. To evaluate the impact of CPAP treatment on erectile dysfunction in OSA patients.

The secondary objectives are:

1. To determine the profile of synthesis of different biomarkers related to endothelial dysfunction and cardiovascular disorder, which are altered as a result of the syndrome of obstructive sleep apnea and its relation to the risk of developing erectile dysfunction.
2. To compare the secretion profile of sex hormones related to control erectile function in a group of patients with syndrome of obstructive sleep apnea with and without erectile dysfunction.
3. To assess the prevalence of erectile dysfunction in patients with OSA.
4. To compare the psychological profile of patients with OSA with and without erectile dysfunction in order to detect psychological distress associated with the risk of developing erectile dysfunction.
5. To evaluate the impact of CPAP treatment on the secretion profile of sex hormones related to control erectile function in OSA patients.
6. To evaluate the impact of CPAP treatment on the psychological profile of patients with erectile disfunction in OSA patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of "obstructive sleep apnea syndrome" (Apnea-Hypopnea Index >10)
* Diagnosis of erectile dysfunction (International Index of Erectile Function score <25)
* Signed informed consent

Exclusion Criteria:

* Psycho-physical inability to perform or collaborate with performing tests.
* Patients presenting any of the following conditions:

  * cardiovascular diseases, neurological diseases (multiple sclerosis, Parkinson's disease, spinal disc disease).
  * history of pelvic or retroperitoneal surgery.
  * congenital or acquired malformations (Peyronie's disease, hypospadias, epispadias, penile fracture).
  * hormonal disorders (hypogonadism, hyperprolactinemia, hyper or hypothyroidism, Cushing's disease).
  * drug addiction and/or alcoholics and treatment with any of the following drugs: antidepressants, antipsychotics.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in International Index Erectile Function (IIEF) score | At baseline and 3 month
  Effect of 3-months CPAP treatment on the changes in the International Index Erectile Function score of patients with Erectile Dysfunction.

SECONDARY OUTCOMES:
Change in Self-Esteem And Relationship (SEAR) score | At baseline and 3 month
  Compare the psychological profile of patients with OSA with and without erectile dysfunction in order to detect psychological distress associated with the risk of developing erectile dysfunction, using SEAR score. Evaluate the impact of CPAP treatment on the change in SEAR score after 3 months.
Changes in Sexual hormone profile (Testosterone, SHBG, free Testosterone, Prolactin, LH, and FSH) | At baseline and 3 month
  Compare the secretion profile of sex hormones related to control erectile function in a group of patients with syndrome of obstructive sleep apnea with and without erectile dysfunction. Evaluate the impact of CPAP treatment on the change in the sexual hormone profile after 3 months. All hormones measured in blood samples by means of Radioimmunoassay.
Changes in Endothelial dysfunction biomarkers (ADMA, ICAM-1, VCAM-1, and VEGF) | At baseline and 3 month
  Determine the profile of synthesis of different biomarkers related to endothelial dysfunction and cardiovascular disorder associated to obstructive sleep apnea and its relation to the risk of developing erectile dysfunction. Evaluate the impact of CPAP treatment on the changes in endothelial dysfunction biomarkers after 3 months. All markers measured in blood samples by means of Radioimmunoassay.

CONTACTS AND LOCATIONS:
Overall Officials: Ferran Barbé, MD, Principal Investigator — Spanish Respiratory Society
Locations (1):
- Hospital Arnau de Vilanova. IRB Lleida. CIBERes, Lleida, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pascual M, de Batlle J, Barbe F, Castro-Grattoni AL, Auguet JM, Pascual L, Vila M, Cortijo A, Sanchez-de-la-Torre M. Erectile dysfunction in obstructive sleep apnea patients: A randomized trial on the effects of Continuous Positive Airway Pressure (CPAP). PLoS One. 2018 Aug 8;13(8):e0201930. doi: 10.1371/journal.pone.0201930. eCollection 2018. PMID 30089160